CLINICAL TRIAL: NCT06348953
Title: Outcome of Bioactive Versus Non-Bioactive System for Restoration of Deep Carious Molars Using Selective Caries Removal Technique: 18 Months Randomized Clinical Trial
Brief Title: Bioactive Versus Non-Bioactive Restorative System in Deep Carious Molars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Ahmed Mohammed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bioactive restorative system
Record Dates: First submitted 2024-03-20; First posted 2024-04-05 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Dental Caries; Dental Diseases; Deep Caries; Tooth Diseases; Tooth Decay; Teeth; Lesion; Caries; Dentin; Dental Restoration Failure of Marginal Integrity; Tooth Demineralization
Keywords: self-etch adhesive; deep caries in permanent molars; bioactive restorative system; selective caries removal; partial caries removal; selective removal to soft caries; bioactive adhesive; bioactive bond; bioactivity; deep carious molars; rct
MeSH Terms: conditions — Dental Caries; Stomatognathic Diseases; Tooth Diseases; Tooth Demineralization

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Conventional non-bioactive restorative system (Comparator) (Active Comparator): deep carious molars restored with conventional resin based restorative system
  Interventions: Other: selective caries removal and conventional non-bioactive restorative system
- Bioactive system (Intervention) (Active Comparator): deep carious molars restored with bioactive resin based restorative system
  Interventions: Other: selective caries removal and bioactive restorative system

INTERVENTIONS:
Other: selective caries removal and conventional non-bioactive restorative system — conventional dental restorative adhesive and resin based composite
  Arms: Conventional non-bioactive restorative system (Comparator)
Other: selective caries removal and bioactive restorative system — bioactive dental restorative resin based system
  Arms: Bioactive system (Intervention)

SUMMARY:
This research study delves into the effectiveness of bioactive and non-bioactive restorative systems in deep carious permanent molars treated with selective caries removal. Selective caries removal techniques aim to preserve as much healthy tooth structure as possible while effectively eliminating carious tissue. The study investigates how the choice of restorative material influences the outcomes of selective caries removal procedures in deep carious lesions. By assessing factors such as restoration integrity, pulpal response, and long-term success rates, the research seeks to provide evidence-based insights into the comparative performance of bioactive and non-bioactive restorative systems in this clinical context.

DETAILED DESCRIPTION:
Deep carious lesions in permanent molars present a significant challenge in restorative dentistry. Traditional approaches to caries removal often involve the removal of excessive healthy tooth structure, leading to weakened teeth and potential pulp exposure. Selective caries removal techniques aim to preserve as much healthy tooth structure as possible while effectively eliminating carious tissue, offering a conservative alternative to traditional methods. In recent years, bioactive restorative materials have emerged as promising alternatives to conventional non-bioactive materials. Bioactive materials are designed to interact with the biological environment, promoting remineralization and potentially enhancing the longevity of restorations. However, limited evidence exists comparing the efficacy of bioactive and non-bioactive restorative systems in deep carious lesions treated with selective caries removal. This study is designed as a prospective, randomized controlled trial. Patients presenting with deep carious lesions in permanent molars will be randomly allocated to receive either a bioactive or non-bioactive restorative system following selective caries removal. Baseline demographic and clinical data will be recorded for each participant. Clinical evaluations will be conducted at regular intervals over a follow-up period of months. Outcome measures will include restoration integrity (e.g retention, marginal adaptation), pulpal response (e.g., sensitivity, vitality).

ELIGIBILITY:
Inclusion Criteria:

* young adult patients (age: 18-40 years) of both genders.
* Able to tolerate necessary restorative procedures.
* Willing to sign the informed consent.
* Accepts the follow-up period.
* Posterior permanent tooth with occlusal proximal deep carious lesion.
* Radiographically (bitewing radiograph) extending to the inner 1/3 of dentine (D3) with a radiopaque layer between the carious lesion and the pulp chamber.
* Sensible teeth according to cold pulp test.

Exclusion criteria:

* Allergy to any restorative materials.
* Patients undergoing orthodontic treatment with fixed appliances.
* Pregnant women.
* Patients with debilitating systemic diseases
* Teeth with previous restorations.
* Spontaneous pain or prolonged pain (more than 15 s) after sensitivity test (cold test), which would indicate irreversible pulpitis.
* Negative sensibility tests, periapical radiolucencies and sensitivity to axial or lateral percussion.
* Mobile teeth, indicating periodontal disease or trauma.
* External or internal resorption.
* Cervical carious lesions.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Biological properties - Post Operative Hypersensitivity and Vitality-Success rate%-Scoring system:Ordinal1-5 | 18 months
  1. excellent(No hypersensitivity,normal vitality
  2. good(Minor hypersensitivity for a limited time,normal vitality
  3. satisfactory(Moderate hypersensitivity-Delayed/mild sensitivity;no subjective complaints,no treatment needed
  4. unsatisfactory(Intense hypersensitivity-Delayed with minor subjective symptoms-No detectable sensitivity-Intervention necessary but not replacement
  5. poor(Intense, acute pulpitis or non-vital tooth-Endodontic treatment is necessary and restoration replacement

SECONDARY OUTCOMES:
Functional properties - (fracture and retention) | 18 months
  1. excelent Frac&Ret:No fractures /Cracks
  2. good Frac&Ret:Small hairline crack
  3. satisfactory Fract and Ret:Two or more or larger hairline cracks and/or material chip fracture not affecting the marginal integrity or approximal contact
  4. unsatisfactory Fract and Ret:Material chip damage marginal quality-approximal contacts-Bulk fracture& partial loss-less than half of restoration
  5. poor Fracture and Retention:(Partial-complete loss of resto. or multiple fractures)
Functional properties - Approximal anatomical form (contact point and contour) | 18 months
  1. excelent Approximal anatomical form (a. contact point b. contour): Normal contact point (floss or 25 μm metal blade can pass) and Normal contour.
  2. good Approximal anatomical form (a. contact point b. contour): Contact slightly too strong but no disadvantage (floss or 25 μm metal blade can only pass with pressure) and slightly deficient contour.
  3. satisfactory Approximal anatomical form: (a. contact point b. contour): Somewhat weak contact, no indication of damage to tooth, gingiva or periodontal structures; 50 μm metal blade can pass and visible deficient contour
  4. unsatisfactory Approximal anatomical form: (a.contact point b.contour)Too weak and possible damage due to food impaction;100 μm metal blade can pass and Inadequate contour (Repairable)
  5. poor Approx. anatomical form (a.contact point b.contour):Too weak and/or clear damage due to food impaction and/or pain/gingivitis with insufficient contour requires replacement.
continue Functional properties (Radiographic Examination -when applicable) | 18 months
  1. excelent xray:No pathology,harmonious transition between restoration &Tooth
  2. good xray:Acceptable material excess present-Positive/negative step present at margin <150 μm
  3. satisfactory xray:Marginal gap<250 μm-Negative steps visible<250 Μm-No adverse effects Noticed-Poor radiopacity of filling
  4. unsatisfactory xray:(Marginal gap >250 μm)(Material excess accessible but not removable)(Negative steps >250μm and reparable)
  5. poor xray:(Secondary caries, large gaps, large overhangs) (Apical pathology) (Fracture/loss of restoration or tooth).
continue Functional properties ( marginal adaptation ) | 18 months
  1. excelent Marginal Adaptation:Harmonious outline,no gaps,white or discolored lines
  2. good Marginal Adaptation:Marginal gap(<150 μm),white line-Small marginal fracture removable by polishing-Slight ditching,slight step/flashes,minor irregularities
  3. satisfactory Marginal Adaptation:Gap<250μm not removable-Several small marginal fractures-Major irregularities,ditching or flash,steps
  4. unsatisfactory Marginal Adapt.:Gap>250μm or dentine/base exposed-Severe ditching or marginal fract. - Larger irregularities or steps -repair necessary
  5. poor Marginal Adaptation:Restoration-complete or partial-is loose but in situ-Generalized major gaps or irregularities.
Biological properties (Recurrence of caries (CAR), erosion, abfraction- Scoring system Ordinal 1-5) | 18 months
  1. = excellent (No secondary or primary caries)
  2. = good (Small and localized 1.Demineralization 2. Erosion or 3. Abfraction)
  3. = satisfactory (Larger areas of 1.Demineralisation 2. Erosion or 3. Abrasion/abfraction, dentine not exposed) (Only preventive measures necessary)
  4. = unsatisfactory (Caries with cavitation and suspected undermining caries) (Erosion in Dentine) (Abrasion/abfraction in dentine) (Localized and accessible can be repaired).
  5. = poor (Deep caries or exposed dentine that is not accessible for repair of restoration)
Success or Failure | 18 months
  Binary Outcome Success (Score 1,2&3) Failure (Score 4 &5)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry - Cairo University, Cairo, Egypt